CLINICAL TRIAL: NCT06395714
Title: Does Performing a Composite Test 3 Months Post-operatively Reduce the Risk of Failure to Return to Sport After Lateral Ankle Ligamentoplasty?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Sport, Bordeaux Mérignac (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-08-SBM_Composite
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Ankle Injuries
Keywords: ligamentoplasty; ankle-go test; sport return
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personnalized physiotherapy (Experimental): Following completion of the ankle go test, patients in "experimental" group will receive specific instructions for continuing their rehabilitation, which will be passed on to the physiotherapist in charge of their rehabilitation.
  These instructions will be adapted according to the results of the composite test and the items identified. The scores of the various functional tests in the composite test will be evaluated to establish the key elements to be taken into account for subsequent management. These instructions will necessarily be personalized according to the scores.
  Interventions: Other: Personnalized physiotherapy
- Usual physiotherapy (Active Comparator): Following completion of the ankle go test, patients in "active comparator" group will undergo conventional rehabilitation following surgery.
  Interventions: Other: Usual physiotherapy

INTERVENTIONS:
Other: Personnalized physiotherapy — Following completion of the ankle go test, patients in "experimental" group will receive specific instructions for continuing their rehabilitation, which will be passed on to the physiotherapist responsible for the rehabilitation.
  Arms: Personnalized physiotherapy
Other: Usual physiotherapy — Following completion of the ankle go test, patients in "active comparator" group will receive usual physiotherapy
  Arms: Usual physiotherapy

SUMMARY:
Ankle sprain is one of the most common pathologies in the general population (between 2.1 and 3.2 per 1000 patients per year). Nearly 40% of patients will develop chronic instability in the year following the sprain. We also know that a premature return to sport is a risk factor for developing chronic instability. However, despite the consensus of experts on the subject which have shown the key physiological elements to evaluate before resuming sport, no test or cohort of tests are proposed to allow a safe return to sport by reducing the risks of relapse. Some very recent studies have appeared on non-operated subjects but this remains a subject that is still too little studied, where the lack of consensus and objective criteria increases the risk of instability. Surgical treatment remains an effective option to reduce the risk of recurrence but failure of the latter can occur in approximately 13-37% of patients depending on the population, due to a relapse or a return to sport which does not correspond to expectations. of the patient.

The objective of the study is therefore to evaluate the predictive nature of a composite test (ANKLE-GO) regarding the return to sport at the same level and the risks of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patient with objective chronic ankle instability who has failed medical treatment and undergone lateral ankle ligament repair surgery
* Patient practicing a sporting activity at least 2 times a week
* Patient able to read, write and understand French
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Minor or over 50 years of age
* Pregnant or breast-feeding patient
* Patient under guardianship, deprived of liberty or under court protection
* Refusal to participate in research
* Patient unable to understand or give informed consent
* Patient having undergone associated surgical procedures modifying the postoperative course
* Patient having undergone revision surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
1-year post-surgery return to sport : Tegner questionnaire | before surgery (anterior practice) and year 1
  evaluation of sport practice level with Tegner questionnaire : Likert scale from 0 (professionnal disability) to 10 (professionnal sport)

SECONDARY OUTCOMES:
Sports level at 1 year post-surgery compared with previous level | Year 1
  Questionnaire "yes/no"
Number of hours of sport per week | before surgery (anterior practice) and year 1
  Self administered questionnaire
Ankle instability scale (FAAM questionnaire : Foot and Ankle Ability Measure) | before surgery (anterior practice) and month 3
  self-administered questionnaire to measure patients' functional progress. It comprises two subscales: a 21-item daily activity subscale, and an 8-item sports subscale. For each subscale, each item is rated on a Likert scale from 0 to 4.
Pain: EVA analog scale | month 1, month 3, month 6, year 1
  EVA scale from 0 (no pain) to 10 (maximal possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Cordier, MD, Principal Investigator — Clinique du sport
Locations (1):
- Clinique du Sport Bordeaux Merignac, Mérignac, France

IPD SHARING:
Plan to Share IPD: No